CLINICAL TRIAL: NCT03592628
Title: Enhancing Postpartum Discharge Instructions for Cesarean Incision Care With Assessment of Comprehension: A Pilot Randomized Controlled Trial
Brief Title: Enhancing Postpartum Discharge Instructions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Rebecca Lawrence, BS (Unknown); Sarah Cohen, MD (Unknown); Rebecca Newbrander, MD (Unknown); Jason K. Baxter, MD (Unknown)
Responsible Party: Principal Investigator, Rebekah McCurdy, Associate Professor, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16D.794
Record Dates: First submitted 2018-07-05; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Health Literacy; Randomized Controlled Trial; Postpartum; Cesarean Delivery Affecting Newborn
MeSH Terms: interventions — Audiovisual Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Instructions (Placebo Comparator): Subjects enrolled in this arm received standardized teach-back regarding discharge instructions as well as the standard printed discharge instructions regarding post-cesarean wound care.
  Interventions: Other: Standard Instructions
- Enhanced Instruction (Experimental): Subjects enrolled in this arm received standardized teach-back regarding discharge instructions as well as the standard printed discharge instructions regarding post-cesarean wound care AND they received an additional printed visual diagram.
  Interventions: Other: Visual Aid

INTERVENTIONS:
Other: Visual Aid — The visual aid was a one-sheet diagram with illustrations of important features of post-cesarean wound care.
  Arms: Enhanced Instruction
Other: Standard Instructions — Standard discharge instructions WITHOUT supplement of visual aid.
  Arms: Standard Instructions

SUMMARY:
Post-cesarean delivery discharge instructions are not currently at an appropriate health literacy level. Enhancing discharge instructions with a visual aid did not improve scores on comprehension quizzes, either immediately or two-weeks post-discharge. However, participants preferred to have access to visual images with discharge instructions.

DETAILED DESCRIPTION:
Objective:

To evaluate the effect of a visual aid on improving comprehension of hospital discharge instructions for cesarean wound care.

Methods:

A randomized control trial with a 1:1 allocation ratio and an intention to treat analysis was performed at an urban, tertiary care center from June-November 2017. Fifty English-speaking patients ages 18-50 who had undergone a cesarean delivery were randomized to receive either standard or enhanced discharge instructions regarding post-cesarean incision care. Enhanced instructions included a visual aid not present in the standard instructions. Participants completed a comprehension quiz prior to hospital discharge and again 2 weeks after discharge as well as the REALM literacy assessment prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent
* Identified as English speaking
* Had a cesarean delivery during the index hospitalization for delivery of their living newborn

Exclusion Criteria:

* Non-English speaking
* Declined to participate
* Required a translator for communication
* Intellectual disability (as self-identified or as determined by healthcare provider)
* Currently incarcerated

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All participants were in-hospital status post a cesarean delivery for delivery of their newborn.
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Comprehension Score Two Weeks Post-Discharge | Two weeks
  Total score on 11-point quiz (Discharge Instructions Comprehension Quiz) administered via phone two weeks post-discharge, score range 1-11 with one point assigned for each correct answer (no subtractions for incorrect answers); higher scores are favorable indicating answers consistent with higher comprehension

SECONDARY OUTCOMES:
Immediate Comprehension | 15 minutes
  Total score on 11-point quiz (Discharge Instructions Comprehension Quiz) administered immediately after discharge instructions reviewed, score range 1-11 with one point assigned for each correct answer (no subtractions for incorrect answers), higher scores are favorable indicating answers consistent with higher comprehension

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah McCurdy, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No